CLINICAL TRIAL: NCT02943785
Title: Edoxaban Versus Standard of Care and Their Effects on Clinical Outcomes in Patients Having Undergone Transcatheter Aortic Valve Implantation (TAVI) - in Atrial Fibrillation
Brief Title: Edoxaban Compared to Standard Care After Heart Valve Replacement Using a Catheter in Patients With Atrial Fibrillation (ENVISAGE-TAVI AF)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Collaborators: Chiltern International Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DU176B-C-U4001; 2016-003930-26 (EudraCT Number)
Record Dates: First submitted 2016-10-21; First posted 2016-10-25 (Estimated); Results first posted 2022-03-24 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Atrial Fibrillation
Keywords: Transcatheter Aortic Valve Implantation -- TAVI; Anticoagulation; Atrial Fibrillation; ENVISAGE-TAVI-AF
MeSH Terms: conditions — Atrial Fibrillation | interventions — edoxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Edoxaban-based Regimen (Experimental): Edoxaban-based regimen 60 mg and 30 mg film coated tablet for once-daily oral use, and 15 mg film coated tablet in case of transitioning at the end of treatment. Dosing must follow the locally approved label.
  Interventions: Drug: Edoxaban-based Regimen
- VKA-based Regimen (Active Comparator): VKA-based regimen oral VKA tablets as selected and provided by the site and used in accordance with the local label. The Investigator will monitor the patient and adjust the VKA dose to maintain the dose within target.
  Interventions: Drug: VKA-based Regimen

INTERVENTIONS:
Drug: Edoxaban-based Regimen — 15 mg, 30 mg and 60 mg film coated tablet for oral use (with anti-platelet therapy pre-declared at randomization if prescribed)
  Other Names: Savaysa; Lixiana
  Arms: Edoxaban-based Regimen
Drug: VKA-based Regimen — Dosed at International Normalized Ratio (INR) levels, which is a test of how long it takes for blood to clot. Standard of Care treatment in the country location (with anti-platelet therapy pre-declared at randomization if prescribed).
  Arms: VKA-based Regimen

SUMMARY:
When the upper chambers of a person's heart receive or generate irregular electrical signals, it causes abnormal rhythm in the heartbeat. This is called atrial fibrillation.

Atrial fibrillation goes along with blood clots that may cause mainly strokes and less often other diseases, such as a heart attack. Some patients with atrial fibrillation have other heart disease, such as heart valves that may need to be replaced using catheters.

Often doctors give patients drugs that reduce those blood clots. These are either vitamin K antagonist (VKA) or direct anticoagulants, such as edoxaban. In these patients, it is unclear which of the drugs is better for reducing stroke without increasing severe bleedings.

DETAILED DESCRIPTION:
Use of Edoxaban in patients with atrial fibrillation (AF) and indication to chronic oral anticoagulation (OAC) after transcatheter aortic valve implantation (TAVI)

Objective:

* To assess the effect of Edoxaban versus vitamin K antagonist (VKA) on net adverse clinical events (NACE), i.e., the composite of all-cause death, myocardial infarction (MI), ischemic stroke, systemic thromboembolism (SEE), valve thrombosis, and major bleeding (International Society on Thrombosis and Haemostasis [ISTH] definition).
* To assess the effect of Edoxaban versus VKA on major bleeding (ISTH definition).

ELIGIBILITY:
Inclusion Criteria:

* Meets protocol-specified criteria for qualification and contraception
* Is willing and able to comply with any restrictions related food, drink and medications
* Voluntarily consents to participate and provides written informed consent prior to any protocol-specific procedures

Exclusion Criteria:

* Has history or current use of over-the-counter medications, dietary supplements, or drugs (including nicotine and alcohol) outside protocol-specified parameters
* Has signs, symptoms or history of any condition that, per protocol or in the opinion of the investigator, might compromise:

  1. the safety or well-being of the participant or study staff
  2. the safety or well-being of the participant's offspring (such as through pregnancy or breast-feeding)
  3. the analysis of results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1426 (Actual)
Dates: Start 2017-03-21 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (230):
- United States (66):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Arizona Sarver Heart Center, Tucson, Arizona
  - Arkansas Site Management Services, Little Rock, Arkansas
  - Loma Linda University Medical Center, Loma Linda, California
  - Cedar-Sinai Heart Institute, Los Angeles, California
  - UCLA Cardiovascular Center, Los Angeles, California
  - University of California - San Francisco, San Francisco, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - Medical Facility Associates, Washington D.C., District of Columbia
  - Cardiology Associate Research, Daytona Beach, Florida
  - International Research Partners, LLC., Doral, Florida
  - Memorial Healthcare Systems, Hollywood, Florida
  - UF Health Jacksonville, Jacksonville, Florida
  - Watson Clinic Center for Research, Lakeland, Florida
  - Tallahassee Research Institute, Inc., Tallahassee, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Carle Foundation Hospital, Urbana, Illinois
  - St. Vincent Heart Center, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Maine Medical Center, Scarborough, Maine
  - Washington Adventist Hospital, Takoma Park, Maryland
  - Baystate Health, Springfield, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Sparrow Clinical Research Institute, Lansing, Michigan
  - MidMichigan Medical Center Midland, Midland, Michigan
  - Michigan Heart, St. Joseph Mercy Health System, Ypsilanti, Michigan
  - Essentia Health, Duluth, Minnesota
  - Mayo Clinic Rochester, Rochester, Minnesota
  - HealthEast Medical Research Institute, Saint Paul, Minnesota
  - Jackson Heart Clinic, Jackson, Mississippi
  - Clinical Investigators LLC, St Louis, Missouri
  - Renown Regional Medical Center, Reno, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - The Valley Hospital, Paramus, New Jersey
  - New Mexico Heart Institute, Albuquerque, New Mexico
  - NY Presbyterian - Brooklyn Methodist Hospital, Brooklyn, New York
  - St. Francis Hospital, East Hills, New York
  - St. Joseph's Physicians, East Syracuse, New York
  - Rochester General Hospital, Geneva, New York
  - Northshore Community Hospital, Manhasset, New York
  - Mt. Sinai Hospital, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Moses H. Cone Memorial Hospital Operating Corporation d/b/a Cone Health, Greensboro, North Carolina
  - East Carolina Heart Institute, Greenville, North Carolina
  - Promedica Toledo Hospital, Toledo, Ohio
  - Oklahoma Heart Hospital Research Foundation, Oklahoma City, Oklahoma
  - Southern Oregon Cardiology, Medford, Oregon
  - Providence Heart and Vascular Institute, Portland, Oregon
  - St. Luke's University Health Network, Bethlehem, Pennsylvania
  - Doylestown Health Cardiothoracic Surgery, Doylestown, Pennsylvania
  - Penn State Health, Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - Pinnacle Health, Wormleysburg, Pennsylvania
  - WellSpan York Hospital, York, Pennsylvania
  - Black Hills Cardiovascular Research, Rapid City, South Dakota
  - SCRI - Centennial Medical Center, Nashville, Tennessee
  - Seton Heart Institute, Austin, Texas
  - Houston Methodist Research Institute, Houston, Texas
  - University of Texas Health Science Center Houston, Houston, Texas
  - Legacy Heart Center, Plano, Texas
  - Inova Heart and Vascular Institute, Falls Church, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - Providence Sacred Heart Medical Research Center, Spokane, Washington
  - CAMC Memorial Hospital, Charleston, West Virginia
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
- Austria (7):
  - Medizinische Universitaet Graz, Graz
  - Clinic Wels-Grieskirchen GmbH, Grieskirchen
  - Universitaetsklinik fuer Innere Medizin III, Innsbruck
  - Klinikum Klagenfurt am Worthersee, Klagenfurt
  - Wilhelminenspital, Vienna
  - Universitätsklinik für Innere Medizin II, Vienna
  - Krankenhaus Hietzing mit Neurologischem Zentrum Rosenhugel, Vienna
- Belgium (8):
  - ASZ Aalst - Aalst campus, Aalst
  - ZNA - Stuivenberg Ziekenhuis Netwerk Antwerpen, Antwerp
  - Hospital Erasme, Brussels
  - UZA - Universtiair Ziekenhuis Antwerpen, Edegem
  - ZOL Genk, Campus Sint-Jan, Genk
  - Jessa Ziekenhuis- Campus Virga Jessa, Hasselt
  - CHU de Liege, Liège
  - AZ Delta Roeselare, Roeselare
- Canada (10):
  - University of Alberta Hospital, Edmonton, Alberta
  - Kingston Health Sciences Centre, Kingston, Ontario
  - London Health Sciences Centre, London, Ontario
  - Newmarket Cardiac Surgery Research Incorporated, Newmarket, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - Hamilton General Hospital, Hamilton
  - Universitè Laval, Québec
  - Horizon Health Network, Saint John
- France (13):
  - CHU d'Angers, Angers
  - Clinique Saint Augustin, Bordeaux
  - Hopital Henri Mondor, Créteil
  - Institut Coeur Poumon - CHRU de Lille, Lille
  - CHU Arnaud de Villeneuve, Montpellier
  - Clinique du Millenaire Service de Cardiologie Interventionelle, Montpellier
  - Institut Mutualiste Montsouris, Paris
  - Hopital Bichat, Paris
  - CHU de Bordeaux Hopital du Haut Leveque, Pessac
  - CHU de Rouen, Rouen
  - Clinique Saint-Hilaire, Rouen
  - Nouvel Hopital Civil, Strasbourg
  - Clinique Pasteur / GCVI, Toulouse
- Germany (29):
  - Kerckhoff-Klinik, Bad Nauheim
  - Herz und Gefaess Klinik, Bad Neustadt an der Saale
  - Segeberger Kliniken, Bad Segeberg
  - Charite Universitatsmedizin Berlin, Berlin
  - Immanuel Klinikum Bernau Herzzentrum Brandenburg, Berlin
  - Gesundheit Nord gGmbH, Bremen
  - Klinikum der Stadt Ludwigshafen, Dortmund
  - St. Johannes - Hospital, Dortmund
  - Heart Center Dresden, University Clinic Technical University Dresden, Dresden
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Elisabeth Krankenhaus Essen Klinik fur Kardiologie und Angiologie, Essen
  - Klinikum Fulda gAG, Fulda
  - Universitatsklinikum Halle (Saale), Halle
  - Asklepios St. Georg Abteilung fuer Kardiologie, Hamburg
  - Heidelberg University Hospital, Heidelberg
  - Universitaetsklinik Schleswig-Holstein Campus Kiel, Kiel
  - MediClin Herzzentrum Lahr/Baden, Lahr
  - Herzzentrum Leipzig, Leipzig
  - Universitatsmedizin Mainz, Zentrum fur Kardiologie, Mainz
  - Deutsches Herzzentrum Munchen, München
  - Universitatsklinikum Essen, Klinik fur Kardiologie, München
  - Klinikum rechts der Isar der Technischen Universitat Munchen, München
  - Klinikum Oldenburg AöR, Oldenburg
  - Uniklinikum Regensburg, Med II, Regensburg
  - Krankenhaus der Barmherzigen, Trier
  - Universitaetsklinikum Tuebingen Medizinische Klinik, Abteilung III, Tübingen
  - Universitatsklinikum Ulm, Ulm
  - Helios Herzzentrum Wuppertal, Wuppertal
  - Universitatsklinikum Wurzburg, Würzburg
- Italy (30):
  - Ospedali Riuniti Torrette Di Ancona, Ancona
  - Policlinico Sant'Orsola-Malpighi, Bologna
  - ASST Spedali Civili di Brescia-UO Cardiologia, Brescia
  - AOU Policlinico Vittorio Emanuele, Catania
  - Magna Graecia University, Catanzaro
  - Ospedale S. Croce e Carle, Cuneo
  - Citta di Lecce Hospital, Lecce
  - Azienda Socio Sanitaria Territoriale di Lecco, Lecco
  - ASST Ovest Milanese - Presidio Ospedallero di Legnana, Legnano
  - Fondazione Toscana Gabriele Monasterio, Massa
  - Ospedale San Raffaele, Milan
  - Centro Cardiologico Monzino IRCCS, Milan
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Clinica Mediterranea, Napoli
  - A.A Dei Colli Monaldi UOC Cardiologia Interventistica, Napoli
  - Azienda Ospedaliera di Padova, Padua
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - IRCCS Policlinico San Matteo, Pavia
  - Centro Cuore Morgagni, Pedara
  - Azienda Ospedaliero-Universitaria Pisana, Pisa
  - IRCCS-ASMN Reggio Emilia, Reggio Emilia
  - AO San Camillo Forlanini, Rome
  - Azienda Ospedaliero-Universitaria Policlinico Umberto I, Rome
  - AOU Careggi, Interventistica Cardiologica Strutturale, Rome
  - Ospedale Sant'Andrea - U.O.S. Emodinamica Cardiologia Interventistica, Rome
  - Istituto Clinico Humanitas, Rozzano
  - AOU S.Giovanni Di Dio e Ruggi D'Aragona, Salerno
  - IRCCS Policlinico San Donato, San Donato Milanese
  - UOC Emodinamica III, Siena
  - Azienda Ospedaliera Integrata di Verona, Verona
- Japan (18):
  - Nagoya Heart Center, Toyohashi, Aichi-ken
  - Kokura Memorial Hospital, Kitakyushu, Fukuoka
  - Ogaki Municipal Hospital, Ōgaki, Gifu
  - Sapporo Higashi Tokushukai Hospital, Sapporo, Hokkaido
  - Tsukuba Medical Center Hospital, Amakubo, Ibaraki
  - Teikyo University Hospital, Tokyo, Itabashi
  - Iwate Medical University Hospital, Morioka, Iwate
  - Tokai University Hospital, Isehara, Kanagawa
  - St. Marianna University School of Medicine Hospital, Kawasaki, Kanagawa
  - Saiseikai Yokohamashi Tobu Hospital, Yokohama, Kanagawa
  - Sendai Kousei Hospital, Sendai, Miyagi
  - Osaka City University Hospital, Abeno Ward, Osaka
  - Kishiwada Tokushukai Hospital, Kishiwada, Osaka
  - Keio University Hospital, Shinjuku, Tokyo
  - Toyohashi Heart Center, Aichi
  - New Tokyo Hospital, Chiba
  - Shonan Kamakura General Hospital, Kanagawa
  - Toyama University Hospital, Toyama
- Netherlands (5):
  - Academic Medical Center, Amsterdam
  - University Medical Center Groningen, Groningen
  - Medisch Centrum Leeuwarden, Leeuwarden
  - Erasmus Medical Center, Rotterdam
  - HagaZiekenhuis, The Hague
- Poland (3):
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Bialystok
  - University Clinical Centre in Gdańsk, Gdansk
  - Szpital Kliniczny Przemienienia Pańskiego Uniwersytetu Medycznego im. Karola Marcinkowskiego w Poznaniu, Poznan
- South Korea (5):
  - Seoul National University Hospital, Seoul, Jongno-gu
  - Seoul St. Mary's Hospital, Seoul, Seocho-gu
  - Yonsei University Severance Hospital, Seoul, Seodaemun-gu
  - Korean University Anam Hospital, Seoul, Seongbuk-gu
  - Asan Medical Center, Seoul, Songpa-gu
- Spain (22):
  - Hospital Universitario Virgen Macarena, Seville, Andalusia
  - Hospital Universitari Germans Trias I Pujol, Badalona, Barcelona
  - Hospital Universitario Donostia, Donostia / San Sebastian, Gipuzkoa
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Complexo Hospitalario Universitario de A Coruna, A Coruña
  - Complexo hospitalario universitario de Santiago de Compostela, A Coruña
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Clinico y Provincial de Barcelona, Barcelona
  - Complejo Asistencial de Granada, Granada
  - Hospital La Luz QuironSalud, Madrid
  - Hospital Universitario La Princesa, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Virgen de la Arrixaca, Murcia
  - Valdecilla Hospital, Santander
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Clinico de Valencia, Valencia
  - Hospital Clinico Universitario de Valladolid, Valladolid
  - Hospital Universitario Alvaro Cunqueiro, Vigo
- Switzerland (4):
  - Universitatsspital Basel, Basel
  - Bern University Hospital, Bern
  - Hopitaux Universitaires de Geneve, Geneva
  - Cardiocentro Ticino, Lugano
- United Kingdom (10):
  - BSUH, Cardiac Research Unit, Brighton, England
  - Papworth Hospital NHS Foundation Trust, Cambridge, England
  - Royal Edinburgh Infirmary, Edinburgh, England
  - Guys St Thomas Hospital, London, England
  - Trent Cardiac Centre, Nottingham, England
  - Oxford University Hospitals, John Radcliffe Hospital, Oxford, England
  - Northern General Hospital, Sheffield, England
  - University Hospital of Wales, Heath Park, Cardiff, Wales
  - University Hospitals of Leicester NHS Trust, Leicester
  - Derriford Hospital, Plymouth

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Van Mieghem NM, Chen C, Hengstenberg C, Van Zyl J, Kimura T, Lang I, Mehran R, Nicolas J, Unverdorben M, Zamorano JL, Dangas GD. Edoxaban Dose Adjustment and Age-Associated Outcomes in Patients With Atrial Fibrillation Post-Transcatheter Aortic Valve Replacement. JACC Adv. 2025 Nov 19;4(12):102329. doi: 10.1016/j.jacadv.2025.102329. Online ahead of print. PMID 41263742
- [Derived] Dangas GD, Unverdorben M, Nicolas J, Hengstenberg C, Chen C, Mollmann H, Jin J, Shawl F, Yamamoto M, Saito S, Hambrecht R, Duggal A, Van Mieghem NM. Comparing Major Gastrointestinal Bleeding in Patients Receiving Edoxaban Versus Warfarin After Transcatheter Aortic Valve Replacement: Results From the Randomized ENVISAGE-TAVI AF Trial. J Am Heart Assoc. 2025 May 20;14(10):e033321. doi: 10.1161/JAHA.123.033321. Epub 2025 May 15. PMID 40371611
- [Derived] Van Mieghem NM, Unverdorben M, Hengstenberg C, Mollmann H, Mehran R, Lopez-Otero D, Nombela-Franco L, Moreno R, Nordbeck P, Thiele H, Lang I, Zamorano JL, Shawl F, Yamamoto M, Watanabe Y, Hayashida K, Hambrecht R, Meincke F, Vranckx P, Jin J, Boersma E, Rodes-Cabau J, Ohlmann P, Capranzano P, Kim HS, Pilgrim T, Anderson R, Baber U, Duggal A, Laeis P, Lanz H, Chen C, Valgimigli M, Veltkamp R, Saito S, Dangas GD; ENVISAGE-TAVI AF Investigators. Edoxaban versus Vitamin K Antagonist for Atrial Fibrillation after TAVR. N Engl J Med. 2021 Dec 2;385(23):2150-2160. doi: 10.1056/NEJMoa2111016. Epub 2021 Aug 28. PMID 34449183
- [Derived] Giacoppo D. Anticoagulation After Transcatheter Aortic Valve Replacement: Evolving Answers and Still Unaddressed Questions. JACC Cardiovasc Interv. 2021 Aug 9;14(15):1714-1716. doi: 10.1016/j.jcin.2021.06.004. Epub 2021 Jul 14. No abstract available. PMID 34274293
- [Derived] Van Mieghem NM, Unverdorben M, Valgimigli M, Mehran R, Boersma E, Baber U, Hengstenberg C, Shi M, Chen C, Saito S, Veltkamp R, Vranckx P, Dangas GD. Edoxaban Versus standard of care and their effects on clinical outcomes in patients having undergone Transcatheter Aortic Valve Implantation in Atrial Fibrillation-Rationale and design of the ENVISAGE-TAVI AF trial. Am Heart J. 2018 Nov;205:63-69. doi: 10.1016/j.ahj.2018.07.006. Epub 2018 Aug 29. PMID 30172099

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1426 participants who met all inclusion criteria and no exclusion criteria were randomized to treatment at 173 clinic sites in Europe, Asia, and North America.
Pre-assignment Details: Participants in the study underwent successful transcatheter aortic valve implantation (TAVI) and had a pre-existing atrial fibrillation (AF) or new onset AF.
Groups:
- Edoxaban: Participants randomized to receive the Edoxaban-based regimen which included 60 mg and 30 mg film coated tablets for once-daily oral use, and 15 mg film coated tablet in case of transitioning at the end of treatment. Dosing followed the locally approved label.
- Vitamin K Antagonist (VKA): Participants randomized to receive the VKA-based regimen which included oral VKA tablets as selected and provided by the site and used in accordance with the local label. The Investigator monitored the patient and adjusted the VKA dose to maintain the dose within target.
Period: Overall Study
Arm/Group | Edoxaban | Vitamin K Antagonist (VKA)
Started | 713 | 713
Completed | 431 | 350
Not Completed | 282 | 363
Not completed — Adverse Event | 112 | 97
Not completed — Withdrawal by Subject | 63 | 126
Not completed — Physician Decision | 23 | 47
Not completed — Death | 46 | 46
Not completed — Lost to Follow-up | 1 | 0
Not completed — Other | 16 | 19
Not completed — Did not receive any study medication | 21 | 28

BASELINE CHARACTERISTICS:
Population: Patient demographics were assessed in the Intent-to-Treat Analysis Set.
Groups:
- Total: Total of all reporting groups
Arm/Group | Edoxaban | Vitamin K Antagonist (VKA) | Total
Number analyzed (Participants) | 713 | 713 | 1426
Age, Continuous [Mean (Standard Deviation); unit: years] | 82.1 (5.4) | 82.1 (5.5) | 82.1 (5.5)
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 5 | 5 | 10
  ≥65 to <75 years | 53 | 55 | 108
  ≥75 to <80 years | 131 | 122 | 253
  ≥80 to <85 years | 289 | 298 | 587
  ≥85 to <90 years | 191 | 183 | 374
  ≥90 years | 44 | 50 | 94
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 347 | 331 | 678
  Male | 366 | 382 | 748
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 92 | 89 | 181
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 4 | 5
  White | 593 | 594 | 1187
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 27 | 26 | 53
Region of Enrollment [Number; unit: participants]
  United States | 77 | 77 | 154
  Japan | 82 | 77 | 159
  United Kingdom | 7 | 10 | 17
  Switzerland | 17 | 17 | 34
  Spain | 172 | 172 | 344
  Canada | 8 | 6 | 14
  Austria | 30 | 32 | 62
  Netherlands | 28 | 27 | 55
  South Korea | 9 | 10 | 19
  Belgium | 17 | 17 | 34
  Poland | 10 | 10 | 20
  Italy | 65 | 67 | 132
  France | 22 | 24 | 46
  Germany | 169 | 167 | 336
Weight [Mean (Standard Deviation); unit: kg] — Population: Baseline characteristics are reported in participants with available baseline data.
  kg
    number analyzed (Participants) | 692 | 685 | 1377
    (all) | 74.6 (17.9) | 76.0 (17.3) | 75.3 (17.6)
Body mass index [Mean (Standard Deviation); unit: kg/m^2] — Population: Baseline characteristics are reported in participants with available baseline data.
  kg/m^2
    number analyzed (Participants) | 691 | 680 | 1371
    (all) | 27.5 (5.7) | 27.9 (5.4) | 27.7 (5.5)
Creatinine Clearance (Cockcroft-Gault formula) [Mean (Standard Deviation); unit: mL/min] — Population: Baseline characteristics are reported in participants with available data.
  mL/min
    number analyzed (Participants) | 692 | 681 | 1373
    (all) | 57.9 (24.0) | 58.6 (24.3) | 58.2 (24.1)
Hypertension [Count of Participants; unit: Participants] | 647 | 657 | 1304
Diabetes mellitus [Count of Participants; unit: Participants] | 270 | 257 | 527
Congestive heart failure [Count of Participants; unit: Participants] — NYHA Class III is defined as participants with cardiac disease producing marked limitation of activity: comfortable at rest. Less than ordinary physical activity causes symptoms. NYHA Class IV is defined as participants with cardiac disease resulting in inability to carry on any physical activity without discomfort. Symptoms may be present even at rest. Participants with NYHA Class III or IV congestive heart disease indicate worse outcome.
  Participants
    Congestive heart failure | 591 | 619 | 1210
    NYHA class III or IV status | 314 | 328 | 642
Mitral valve disease [Count of Participants; unit: Participants] | 57 | 60 | 117
History of stroke or transient ischemic attack [Count of Participants; unit: Participants] | 123 | 116 | 239
Coronary artery disease [Count of Participants; unit: Participants]
  History of coronary artery disease | 293 | 297 | 590
  Prior coronary bypass surgery | 67 | 60 | 127
  Prior percutaneous coronary intervention | 176 | 192 | 368
  Prior myocardial infarction | 97 | 101 | 198

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Net Adverse Clinical Events (Adjudicated Data) Based on ISTH Criteria in Participants Taking Edoxaban vs VKA
Description: The composite endpoint net adverse clinical events (NACE) included all-cause death, myocardial infarction (MI), ischemic stroke, systemic embolic events (SEE), valve thrombosis, and major bleeding per definition of the International Society on Thrombosis and Haemostasis (ISTH].
Time Frame: Baseline through study completion, up to 36 months post-dose
Population: Net adverse clinical events were assessed in the Intent-to-Treat (ITT) Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Edoxaban | Vitamin K Antagonist (VKA)
Number analyzed (Participants) | 713 | 713
Participants | 170 | 157
Statistical Analysis 1: Comparison: Edoxaban vs Vitamin K Antagonist (VKA); Test type: Non-Inferiority — The two-sided p-value (Noninferiority) was based on the noninferiority margin of 1.38; p = 0.0141, Regression, Cox; Cox Proportional Hazard = 1.05, 95% CI 2-sided [0.85 to 1.31]

2. Primary Outcome: Number of Participants Who Experienced Major Bleeding (Adjudicated Data) Based on ISTH Criteria in Participants Taking Edoxaban vs VKA
Description: ISTH Bleeding Criteria for Major Bleeding are defined as clinically overt bleeding that is associated with: a fall in hemoglobin of 2 g/dL (1.24 mmol/L) or more, or a transfusion of 2 or more units of whole blood or packed red blood cells, or symptomatic bleeding into a critical site or organ such as intracranial, intraspinal, intraocular, retroperitoneal, pericardial, intra-articular, or intramuscular with compartment syndrome, or a fatal outcome.
Time Frame: Baseline through study completion, up to 36 months post-dose
Population: Bleeding events were assessed in the ITT Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Edoxaban | Vitamin K Antagonist (VKA)
Number analyzed (Participants) | 713 | 713
Participants | 98 | 68
Statistical Analysis 1: Comparison: Edoxaban vs Vitamin K Antagonist (VKA); Test type: Non-Inferiority — The two-sided p-value (Noninferiority) was based on the noninferiority margin of 1.38; p = 0.9267, Regression, Cox; Cox Proportional Hazard = 1.40, 95% CI 2-sided [1.03 to 1.91]

3. Secondary Outcome: Number of Participants Who Experienced Net Adverse Clinical Events (Adjudicated Data) Based on TIMI Criteria in Participants Taking Edoxaban vs VKA
Description: The composite endpoint of net adverse event clinical events (NACE) included all-cause death, myocardial infarction (MI), ischemic stroke, systemic embolic events (SEE), valve thrombosis, and major bleeding based on Thrombolysis in Myocardial Infarction (TIMI) criteria. Bleeding by TIMI criteria was defined as the following: (1) Major, any intracranial hemorrhage or any clinically overt bleeding, (including bleeding evident in imaging studies) associated with a fall of hemoglobin (Hb) of ≥ 5g/dL or fatal bleeding and (2) Minor, any clinically overt bleeding associated with a fall in Hb ≥ 3g/dL but < 5 g/dL.
Time Frame: Baseline through study completion, up to 36 months post-dose
Population: Net adverse clinical events were assessed in the ITT Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Edoxaban | Vitamin K Antagonist (VKA)
Number analyzed (Participants) | 713 | 713
Participants
  Composite endpoint NACE (TIMI) | 154 | 141
  Composite of major and minor bleeding (TIMI) | 72 | 42

4. Secondary Outcome: Number of Participants Who Experienced Net Adverse Clinical Events (Adjudicated Data) Based on BARC Type 3 or 5 Criteria in Participants Taking Edoxaban vs VKA
Description: The composite endpoint of net adverse event clinical events (NACE) included all-cause death, MI, ischemic stroke, SEE, valve thrombosis, and major bleeding based on Bleeding Academic Research Consortium (BARC) Type 3 or 5 criteria. Major bleeding by BARC criteria was defined as Type 3: clinical, laboratory, and/or imaging evidence of bleeding with provider responses; Type 3a: any transfusion with overt bleeding; overt bleeding plus Hb drop of 3 to < 5 g/dL; Type 3b: overt bleeding plus Hb drop ≥ 5 g/dL; cardiac tamponade; bleeding requiring surgical intervention; bleeding requiring intravenous vasoactive drugs; Type 3c: intracranial hemorrhage; subcategories confirmed by autopsy, imaging, or lumbar puncture; intraocular bleed compromising vision; Type 5: fatal bleeding; Type 5a: probable fatal bleeding; no autopsy or imaging confirmation but clinically suspicious; Type 5b: definite fatal bleeding; overt bleeding or autopsy or imaging confirmation
Time Frame: Baseline through study completion, up to 36 months post-dose
Population: Net adverse clinical events were assessed in the ITT Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Edoxaban | Vitamin K Antagonist (VKA)
Number analyzed (Participants) | 713 | 713
Participants
  Composite endpoint NACE (BARC Type 3 or 5) | 164 | 151
  Major bleeding (BARC Type 3 or 5) | 89 | 57

5. Secondary Outcome: Number of Participants Who Experienced Net Adverse Clinical Events (Adjudicated Data) Based on GUSTO Criteria in Participants Taking Edoxaban vs VKA
Description: The composite endpoint of net adverse event clinical events (NACE) included all-cause death, MI, ischemic stroke, SEE, valve thrombosis, and major bleeding based on Global Utilization of Streptokinase and Tissue Plasminogen Activator for Occluded Coronary Arteries (GUSTO). GUSTO criteria was defined as the following: severe or life threatening: intracerebral hemorrhage or resulting in substantial hemodynamic compromise requiring treatment and moderate: requiring blood transfusion but not resulting in hemodynamic compromise.
Time Frame: Baseline through study completion, up to 36 months post-dose
Population: Net adverse clinical events were assessed in the ITT Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Edoxaban | Vitamin K Antagonist (VKA)
Number analyzed (Participants) | 713 | 713
Participants
  Composite endpoint NACE (GUSTO) | 160 | 146
  Severe or life threatening and moderate bleeding (GUSTO) | 82 | 51

6. Secondary Outcome: Number of Participants Who Experienced Major Adverse Cardiac Events (MACE) in Participants Taking Edoxaban vs VKA (Adjudicated Data)
Description: Major adverse cardiac events (MACE) is defined as the composite of all-cause death (excluding adjudicated non-cardiac death), MI, or repeat coronary revascularization of the target lesion.
Time Frame: Baseline through study completion, up to 36 months post-dose
Population: MACE were assessed in the ITT Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Edoxaban | Vitamin K Antagonist (VKA)
Number analyzed (Participants) | 713 | 713
Participants | 61 | 53

7. Secondary Outcome: Number of Participants Who Experienced Major Adverse Cardiac and Cerebrovascular Events (MACCE) in Participants Taking Edoxaban vs VKA (Adjudicated Data)
Description: Major adverse cardiac and cerebrovascular events (MACCE) is defined as the composite of all-cause death (excluding adjudicated non-cardiac death), MI, stroke (ischemic, hemorrhagic, or undetermined), or repeat coronary revascularization of the target lesion
Time Frame: Baseline through study completion, up to 36 months post-dose
Population: MACE were assessed in the ITT Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Edoxaban | Vitamin K Antagonist (VKA)
Number analyzed (Participants) | 713 | 713
Participants | 86 | 80

8. Secondary Outcome: Number of Participants Who Experienced a Composite of Adverse Events in Participants Taking Edoxaban vs VKA (Adjudicated Data)
Description: A composite of clinical adverse events included cardiovascular death, MI ischemic stroke, SEE, valve thrombosis, and major bleeding as defined by ISTH criteria.
Time Frame: Baseline through study completion, up to 36 months post-dose
Population: A composite of adverse events was assessed in the ITT Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Edoxaban | Vitamin K Antagonist (VKA)
Number analyzed (Participants) | 713 | 713
Participants | 151 | 123

9. Secondary Outcome: Number of Participants Who Experienced Stroke Events (Ischemic, Hemorrhagic, Undetermined) in Participants Taking Edoxaban vs VKA (Adjudicated Data)
Description: Stroke events are categorized as any stroke, fatal stroke, and non-fatal stroke.
Time Frame: Baseline through study completion, up to 36 months post-dose
Population: Stroke events were assessed in the ITT Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Edoxaban | Vitamin K Antagonist (VKA)
Number analyzed (Participants) | 713 | 713
Participants
  Any stroke (ischemic, hemorrhagic, or undetermined) | 29 | 35
  Fatal stroke (ischemic, hemorrhagic, or undetermined) | 4 | 3
  Non-fatal stroke (ischemic, hemorrhagic, or undetermined) | 25 | 32

10. Secondary Outcome: Number of Participants Who Experienced Systemic Embolic Events in Participants Taking Edoxaban vs VKA (Adjudicated Data)
Description: Systemic thromboembolism [non-central nervous system] is defined as abrupt vascular insufficiency of an extremity or organ associated with clinical or radiological evidence of arterial occlusion in the absence of other likely mechanisms, (e.g., trauma, atherosclerosis, instrumentation).
Time Frame: Baseline through study completion, up to 36 months post-dose
Population: Systemic embolic events (SEE) were assessed in the ITT Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Edoxaban | Vitamin K Antagonist (VKA)
Number analyzed (Participants) | 713 | 713
Participants | 2 | 3

11. Secondary Outcome: Number of Participants Who Experienced Myocardial Infarctions (MI) in Participants Taking Edoxaban vs VKA (Adjudicated Data)
Description: Peri-procedural MI was defined as new ischemic symptoms or signs and elevated cardiac biomarkers within 72 hours after index procedure, consisting of at least one sample post-procedure with a peak value exceeding 15x as the upper reference limit (URL) for troponin or 5x for CK-MB. Spontaneous MI is defined as any one of the following: Detection of rise and/or fall of cardiac biomarkers with at least one value above the 99th percentile URL, together with the evidence of myocardial ischemia with at least one of the following: Symptoms of ischemia; ECG changes indicative of new ischemia; New pathological Q-waves in at least two contiguous leads; Imaging evidence of a new loss of viable myocardium or new wall motion abnormality; Sudden, unexpected cardiac death, involving cardiac arrest, often with symptoms suggestive of myocardial ischemia, and accompanied by new ST elevation or new left bundle branch block, and/or evidence of fresh thrombus; Pathological findings of an acute MI.
Time Frame: Baseline through study completion, up to 36 months post-dose
Population: Myocardial infarctions were assessed in the ITT Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Edoxaban | Vitamin K Antagonist (VKA)
Number analyzed (Participants) | 713 | 713
Participants | 12 | 7

12. Secondary Outcome: Number of Participants Who Experienced Valve Thrombosis in Participants Taking Edoxaban vs VKA (Adjudicated Data)
Description: Valve thrombosis was defined as any thrombus attached to or near an implanted valve that occludes part of the blood flow path, interferes with valve function, or is sufficiently large to warrant treatment.
Time Frame: Baseline through study completion, up to 36 months post-dose
Population: Valve thrombosis were assessed in the ITT Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Edoxaban | Vitamin K Antagonist (VKA)
Number analyzed (Participants) | 713 | 713
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were collected from the Safety Analysis Set from baseline up 4 weeks post-discontinuation of study treatment or through study completion, up to 36 months post-dose.
Description: Treatment-emergent adverse events are defined as events which start on or after any first dose of the assigned study medication regimen or started prior to but then worsened after any first dose of the assigned study medication regimen.
Groups:
- Edoxaban: Participants randomized to receive the Edoxaban-based regimen which included 60 mg and 30 mg film coated tablet for once-daily oral use, and 15 mg film coated tablet in case of transitioning at the end of treatment. Dosing followed the locally approved label.
Arm/Group | Edoxaban | Vitamin K Antagonist (VKA)
All-Cause Mortality (participants affected / at risk) | 83/693 | 78/684
Serious Adverse Events (participants affected / at risk) | 388/693 | 372/684
Other Adverse Events (participants affected / at risk) | 522/693 | 429/684
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Edoxaban (N=693) | Vitamin K Antagonist (VKA) (N=684)
Pneumonia (Infections and infestations) | 39 | 37
Urinary tract infection (Infections and infestations) | 21 | 17
Endocarditis (Infections and infestations) | 14 | 7
Respiratory tract infection (Infections and infestations) | 7 | 13
Sepsis (Infections and infestations) | 6 | 7
Bronchitis (Infections and infestations) | 4 | 5
COVID-19 (Infections and infestations) | 2 | 6
Septic shock (Infections and infestations) | 5 | 3
Urosepsis (Infections and infestations) | 6 | 2
Cellulitis (Infections and infestations) | 3 | 4
Gastroenteritis (Infections and infestations) | 3 | 3
Bacteraemia (Infections and infestations) | 2 | 3
COVID-19 pneumonia (Infections and infestations) | 1 | 4
Influenza (Infections and infestations) | 4 | 1
Enterococcal sepsis (Infections and infestations) | 2 | 2
Lower respiratory tract infection (Infections and infestations) | 3 | 1
Appendicitis (Infections and infestations) | 0 | 3
Cystitis (Infections and infestations) | 3 | 0
Erysipelas (Infections and infestations) | 3 | 0
Infection (Infections and infestations) | 1 | 2
Intervertebral discitis (Infections and infestations) | 1 | 2
Staphylococcal bacteraemia (Infections and infestations) | 2 | 1
Staphylococcal sepsis (Infections and infestations) | 2 | 1
Streptococcal endocarditis (Infections and infestations) | 3 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 1
Endocarditis staphylococcal (Infections and infestations) | 1 | 1
Enterococcal bacteraemia (Infections and infestations) | 1 | 1
Enterococcal infection (Infections and infestations) | 0 | 2
Epididymitis (Infections and infestations) | 1 | 1
Escherichia sepsis (Infections and infestations) | 2 | 0
Gangrene (Infections and infestations) | 1 | 1
Herpes zoster (Infections and infestations) | 2 | 0
Klebsiella infection (Infections and infestations) | 1 | 1
Pulmonary sepsis (Infections and infestations) | 1 | 1
Pyelonephritis (Infections and infestations) | 1 | 1
Streptococcal bacteraemia (Infections and infestations) | 1 | 1
Abscess soft tissue (Infections and infestations) | 1 | 0
Acinetobacter bacteraemia (Infections and infestations) | 1 | 0
Alveolar osteitis (Infections and infestations) | 1 | 0
Anal abscess (Infections and infestations) | 0 | 1
Aspergilloma (Infections and infestations) | 0 | 1
Bacterial sepsis (Infections and infestations) | 1 | 0
Citrobacter sepsis (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Cystitis klebsiella (Infections and infestations) | 1 | 0
Device-related sepsis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Endocarditis enterococcal (Infections and infestations) | 1 | 0
Escherichia bacteraemia (Infections and infestations) | 1 | 0
Escherichia infection (Infections and infestations) | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0
Fracture infection (Infections and infestations) | 1 | 0
Fungal tracheitis (Infections and infestations) | 0 | 1
Gastric infection (Infections and infestations) | 0 | 1
Groin infection (Infections and infestations) | 0 | 1
Herpes zoster oticus (Infections and infestations) | 1 | 0
Infected lymphocele (Infections and infestations) | 0 | 1
Infective aneurysm (Infections and infestations) | 0 | 1
Klebsiella bacteraemia (Infections and infestations) | 1 | 0
Klebsiella sepsis (Infections and infestations) | 0 | 1
Medical device site infection (Infections and infestations) | 0 | 1
Mycotic corneal ulcer (Infections and infestations) | 1 | 0
Nosocomial infection (Infections and infestations) | 1 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 0 | 1
Pneumococcal bacteraemia (Infections and infestations) | 0 | 1
Pneumococcal sepsis (Infections and infestations) | 1 | 0
Pneumonia pneumococcal (Infections and infestations) | 0 | 1
Pneumonia streptococcal (Infections and infestations) | 0 | 1
Postoperative wound infection (Infections and infestations) | 0 | 1
Pseudomonal sepsis (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 1
Respiratory tract infection viral (Infections and infestations) | 1 | 0
Rhinovirus infection (Infections and infestations) | 1 | 0
Salmonellosis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Streptococcal sepsis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chronic myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to pelvis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Myeloproliferative neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Refractory cytopenia with unilineage dysplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ureteric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 31 | 11
Blood loss anaemia (Blood and lymphatic system disorders) | 5 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 3 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 6
Anaemia folate deficiency (Blood and lymphatic system disorders) | 2 | 0
Hypochromic anaemia (Blood and lymphatic system disorders) | 2 | 0
Normocytic anaemia (Blood and lymphatic system disorders) | 2 | 0
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 1 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Nephrogenic anaemia (Blood and lymphatic system disorders) | 1 | 0
Normochromic anaemia (Blood and lymphatic system disorders) | 1 | 0
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Splenic infarction (Blood and lymphatic system disorders) | 1 | 0
Spontaneous haematoma (Blood and lymphatic system disorders) | 0 | 1
Anaphylatic shock (Immune system disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 3 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 3
Fluid overload (Metabolism and nutrition disorders) | 2 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 2
Cachexia (Metabolism and nutrition disorders) | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 2
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 1
Acidosis (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 | 0
Fluid retention (Metabolism and nutrition disorders) | 1 | 0
Fructose intolerance (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 4 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Drug dependence (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1
Stress (Psychiatric disorders) | 0 | 1
Syncope (Nervous system disorders) | 13 | 12
Ischaemic stroke (Nervous system disorders) | 9 | 10
Transient ischaemic attack (Nervous system disorders) | 7 | 8
Dizziness (Nervous system disorders) | 6 | 5
Cerebral haemorrhage (Nervous system disorders) | 5 | 1
Cerebral infarction (Nervous system disorders) | 2 | 4
Embolic stroke (Nervous system disorders) | 4 | 1
Cognitive disorder (Nervous system disorders) | 3 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 3
Haemorrhage stroke (Nervous system disorders) | 1 | 3
Chorea (Nervous system disorders) | 2 | 1
Epilepsy (Nervous system disorders) | 3 | 0
Loss of consciousness (Nervous system disorders) | 3 | 0
Presyncope (Nervous system disorders) | 1 | 2
Cerebral ischaemia (Nervous system disorders) | 2 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 2
Dementia (Nervous system disorders) | 1 | 1
Embolic cerebral infarction (Nervous system disorders) | 1 | 1
Lacunar infarction (Nervous system disorders) | 2 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 1
Altered state of consciousness (Nervous system disorders) | 0 | 1
Amnesia (Nervous system disorders) | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0
Central nervous system lesion (Nervous system disorders) | 1 | 0
Cerebellar infarction (Nervous system disorders) | 0 | 1
Cerebral microangiopathy (Nervous system disorders) | 0 | 1
Cerebrovascular disorder (Nervous system disorders) | 0 | 1
Choreoathetosis (Nervous system disorders) | 1 | 0
Cubital tunnel syndrome (Nervous system disorders) | 1 | 0
Dementia Alzheimer's type (Nervous system disorders) | 0 | 1
Dysaesthesia (Nervous system disorders) | 0 | 1
Dysarthria (Nervous system disorders) | 1 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Hypertensive encephalopathy (Nervous system disorders) | 1 | 0
Intraventricular haemorrhage (Nervous system disorders) | 1 | 0
Lacunar stroke (Nervous system disorders) | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Parkinson's disease (Nervous system disorders) | 1 | 0
Partial seizures (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 1 | 0
Status epileticus (Nervous system disorders) | 1 | 0
Vascular encephalopathy (Nervous system disorders) | 1 | 0
Cataract (Eye disorders) | 2 | 1
Retinal artery occlusion (Eye disorders) | 2 | 1
Amaurosis fugax (Eye disorders) | 0 | 1
Choroidal detachment (Eye disorders) | 1 | 0
Retinal haemorrhage (Eye disorders) | 0 | 1
Vitreous detachment (Eye disorders) | 1 | 0
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 | 0
Vestibular disorder (Ear and labyrinth disorders) | 0 | 1
Vestibular paroxysmia (Ear and labyrinth disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 57 | 64
Atrial fibrillation (Cardiac disorders) | 17 | 18
Cardiac failure congestive (Cardiac disorders) | 23 | 12
Cardiac failure acute (Cardiac disorders) | 8 | 11
Atrioventricular block complete (Cardiac disorders) | 9 | 6
Mitral valve incompetence (Cardiac disorders) | 6 | 8
Bradycardia (Cardiac disorders) | 6 | 3
Cardiac arrest (Cardiac disorders) | 2 | 7
Atrial flutter (Cardiac disorders) | 6 | 1
Acute myocardial infarction (Cardiac disorders) | 4 | 2
Angina pectoris (Cardiac disorders) | 2 | 4
Sinus node dysfunction (Cardiac disorders) | 4 | 2
Pericardial effusion (Cardiac disorders) | 4 | 1
Tachyarrhythmia (Cardiac disorders) | 2 | 3
Atrioventricular block (Cardiac disorders) | 3 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 4
Ventricular tachycardia (Cardiac disorders) | 2 | 2
Bundle branch block left (Cardiac disorders) | 2 | 1
Cardiac failure chronic (Cardiac disorders) | 1 | 2
Coronary artery disease (Cardiac disorders) | 3 | 0
Aortic valve stenosis (Cardiac disorders) | 2 | 0
Arrhythmia (Cardiac disorders) | 1 | 1
Cardiac asthma (Cardiac disorders) | 1 | 1
Cardiac tamponade (Cardiac disorders) | 1 | 1
Cardiopulmonary failure (Cardiac disorders) | 2 | 0
Left ventricular failure (Cardiac disorders) | 2 | 0
Myocardial infarction (Cardiac disorders) | 0 | 2
Sinus arrest (Cardiac disorders) | 1 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Acute left ventricular failure (Cardiac disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 1
Aortic valve disease (Cardiac disorders) | 0 | 1
Aortic valve incompetence (Cardiac disorders) | 0 | 1
Atrial tachycardia (Cardiac disorders) | 1 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 1
Atrioventricular block second degree (Cardiac disorders) | 1 | 0
Bifascicular block (Cardiac disorders) | 1 | 0
Bradyarrhythmia (Cardiac disorders) | 1 | 0
Cardiogenic shock (Cardiac disorders) | 0 | 1
Cardiorenal syndrome (Cardiac disorders) | 0 | 1
Chronic left ventricular failure (Cardiac disorders) | 0 | 1
Conduction disorder (Cardiac disorders) | 1 | 0
Cor pulmonale (Cardiac disorders) | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 1
Intracardiac thrombus (Cardiac disorders) | 1 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 0
Mitral valve disease (Cardiac disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 1 | 0
Prosthetic cardiac valve thrombosis (Cardiac disorders) | 1 | 0
Right ventricular failure (Cardiac disorders) | 0 | 1
Stress cardiomyopathy (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Ventricular dysfunction (Cardiac disorders) | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 7 | 5
Haematoma (Vascular disorders) | 2 | 9
Hypertensive crisis (Vascular disorders) | 8 | 1
Orthostatic hypotension (Vascular disorders) | 3 | 1
Hypertension (Vascular disorders) | 2 | 1
Aortic dissection (Vascular disorders) | 2 | 0
Circulatory collapse (Vascular disorders) | 0 | 2
Hypotension (Vascular disorders) | 2 | 0
Iliac artery stenosis (Vascular disorders) | 2 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 2
Phlebitis (Vascular disorders) | 1 | 1
Aortic aneurysm (Vascular disorders) | 1 | 0
Aortic occlusion (Vascular disorders) | 1 | 0
Aortic perforation (Vascular disorders) | 1 | 0
Aortic thrombosis (Vascular disorders) | 1 | 0
Arterial haemorrhage (Vascular disorders) | 1 | 0
Arterial occlusive disease (Vascular disorders) | 0 | 1
Arteriovenous fistula (Vascular disorders) | 0 | 1
Blue toe syndrome (Vascular disorders) | 1 | 0
Diabetic vascular disorder (Vascular disorders) | 0 | 1
Extremity necrosis (Vascular disorders) | 1 | 0
Femoral artery embolism (Vascular disorders) | 0 | 1
Haemorrhage (Vascular disorders) | 0 | 1
Hypovolaemic shock (Vascular disorders) | 0 | 1
Peripheral artery aneurysm (Vascular disorders) | 1 | 0
Peripheral artery thrombosis (Vascular disorders) | 0 | 1
Peripheral embolism (Vascular disorders) | 0 | 1
Peripheral vascular disorder (Vascular disorders) | 1 | 0
Peripheral venous disease (Vascular disorders) | 0 | 1
Shock haemorrhagic (Vascular disorders) | 0 | 1
Subclavian vein thrombosis (Vascular disorders) | 1 | 0
Varicose vein (Vascular disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 | 8
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7 | 8
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 5 | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 | 3
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngeal haematoma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pickwickian syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 16 | 7
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 8 | 4
Diarrhoea (Gastrointestinal disorders) | 7 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 5 | 3
Inguinal hernia (Gastrointestinal disorders) | 2 | 6
Rectal haemorrhage (Gastrointestinal disorders) | 4 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Anal haemorrhage (Gastrointestinal disorders) | 3 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 2
Intestinal obstruction (Gastrointestinal disorders) | 2 | 1
Melaena (Gastrointestinal disorders) | 3 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Diverticulum intestinal hemorrhagic (Gastrointestinal disorders) | 2 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2
Abdominal hernia (Gastrointestinal disorders) | 0 | 1
Anal fissure (Gastrointestinal disorders) | 1 | 0
Chronic gastritis (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 0
Enterocele (Gastrointestinal disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastric perforation (Gastrointestinal disorders) | 0 | 1
Gastric polyps (Gastrointestinal disorders) | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastroduodenal ulcer (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Intestinal polyp (Gastrointestinal disorders) | 1 | 0
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 | 0
Mechanical ileus (Gastrointestinal disorders) | 0 | 1
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 0
Pancreatic failure (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Pancreatitis necrotising (Gastrointestinal disorders) | 0 | 1
Subileus (Gastrointestinal disorders) | 0 | 1
Ulcerative duodenitis (Gastrointestinal disorders) | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 4 | 2
Cholelithiasis (Hepatobiliary disorders) | 2 | 2
Cholangitis (Hepatobiliary disorders) | 2 | 0
Cholangitis acute (Hepatobiliary disorders) | 0 | 2
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 3
Diabetic foot (Skin and subcutaneous tissue disorders) | 2 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer haemorrhage (Skin and subcutaneous tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 5 | 3
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Chest wall haematoma (Musculoskeletal and connective tissue disorders) | 0 | 1
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 | 1
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Soft tissue disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 18 | 17
Haematuria (Renal and urinary disorders) | 11 | 3
Chronic kidney disease (Renal and urinary disorders) | 1 | 5
Renal failure (Renal and urinary disorders) | 4 | 2
Urinary retention (Renal and urinary disorders) | 4 | 0
End stage renal disease (Renal and urinary disorders) | 0 | 2
Nephrolithiasis (Renal and urinary disorders) | 1 | 1
Renal impairment (Renal and urinary disorders) | 1 | 1
Calculus bladder (Renal and urinary disorders) | 1 | 0
Renal haematoma (Renal and urinary disorders) | 1 | 0
Renal infarct (Renal and urinary disorders) | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 1
Urethral haemorrhage (Renal and urinary disorders) | 1 | 0
Urethral stenosis (Renal and urinary disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 1
Female genital tract fistula (Reproductive system and breast disorders) | 1 | 0
Pelvic haematoma (Reproductive system and breast disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Rectocele (Reproductive system and breast disorders) | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Death (General disorders) | 8 | 3
General physical health deterioration (General disorders) | 3 | 6
Asthenia (General disorders) | 4 | 4
Multiple organ dysfunction syndrome (General disorders) | 5 | 2
Non-cardiac chest pain (General disorders) | 4 | 2
Sudden death (General disorders) | 4 | 2
Impaired healing (General disorders) | 1 | 2
Pyrexia (General disorders) | 3 | 0
Malaise (General disorders) | 1 | 1
Oedema peripheral (General disorders) | 1 | 1
Pacemaker generated arrhythmia (General disorders) | 2 | 0
Chest discomfort (General disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Injection site haematoma (General disorders) | 0 | 1
Peripheral swelling (General disorders) | 0 | 1
Stent-graft endoleak (General disorders) | 0 | 1
Sudden cardiac death (General disorders) | 0 | 1
Systemic inflammatory response syndrome (General disorders) | 1 | 0
International normalised ratio increased (Investigations) | 1 | 5
Haemoglobin decreased (Investigations) | 2 | 0
Troponin increased (Investigations) | 1 | 1
Anticoagulation drug level above therapeutic (Investigations) | 0 | 1
Blood lactic acid increased (Investigations) | 1 | 0
Coronavirus test positive (Investigations) | 1 | 0
Ejection fraction decreased (Investigations) | 0 | 1
General physical condition normal (Investigations) | 0 | 1
Heart rate irregular (General disorders) | 0 | 1
Hepatic enzyme increased (General disorders) | 1 | 0
Inflammatory marker increased (General disorders) | 1 | 0
Myocardial necrosis marker increased (General disorders) | 0 | 1
Weight increased (General disorders) | 0 | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 6 | 8
Fall (Injury, poisoning and procedural complications) | 9 | 4
Femur fracture (Injury, poisoning and procedural complications) | 5 | 6
Subdural haematoma (Injury, poisoning and procedural complications) | 3 | 5
Femoral neck fracture (Injury, poisoning and procedural complications) | 4 | 3
Head injury (Injury, poisoning and procedural complications) | 3 | 3
Hip fracture (Injury, poisoning and procedural complications) | 2 | 4
Pelvic fracture (Injury, poisoning and procedural complications) | 2 | 4
Humerus fracture (Injury, poisoning and procedural complications) | 2 | 3
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 4
Spinal compression fracture (Injury, poisoning and procedural complications) | 2 | 2
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 2 | 2
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 | 3
Ankle fracture (Injury, poisoning and procedural complications) | 2 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 3 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 3
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 1
Radius fracture (Injury, poisoning and procedural complications) | 2 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 1
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 | 2
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 1
Vascular access site pseduoaneurysm (Injury, poisoning and procedural complications) | 1 | 1
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 | 1
Bone contusion (Injury, poisoning and procedural complications) | 1 | 0
Chest injury (Injury, poisoning and procedural complications) | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1
Colon injury (Injury, poisoning and procedural complications) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0
Extradural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Face injury (Injury, poisoning and procedural complications) | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0
Foreign body in gastrointestinal tract (Injury, poisoning and procedural complications) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Fractured sacrum (Injury, poisoning and procedural complications) | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1
Heat illness (Injury, poisoning and procedural complications) | 1 | 0
Heat stroke (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Open globe injury (Injury, poisoning and procedural complications) | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Post procedural fever (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Postoperative delirium (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Seroma (Injury, poisoning and procedural complications) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1
Vascular access site haematoma (Injury, poisoning and procedural complications) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
Device leakage (Product Issues) | 3 | 0
Device malfunction (Product Issues) | 1 | 1
Device power source issue (Product Issues) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Edoxaban (N=693) | Vitamin K Antagonist (VKA) (N=684)
Urinary tract infection (Infections and infestations) | 63 | 45
Pneumonia (Infections and infestations) | 45 | 43
Anaemia (Blood and lymphatic system disorders) | 62 | 40
Dizziness (Nervous system disorders) | 47 | 33
Cardiac failure (Cardiac disorders) | 78 | 85
Atrial fibrillation (Cardiac disorders) | 23 | 36
Haematoma (Vascular disorders) | 26 | 41
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 64 | 30
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 39 | 35
Haematuria (Renal and urinary disorders) | 40 | 18
Fall (Injury, poisoning and procedural complications) | 35 | 23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-29): https://cdn.clinicaltrials.gov/large-docs/85/NCT02943785/Prot_SAP_000.pdf